CLINICAL TRIAL: NCT01693783
Title: A Phase 2 Study of Ipilimumab in Women With Metastatic or Recurrent HPV-Related Cervical Carcinoma of Either Squamous Cell or Adenocarcinoma Histologies
Brief Title: Ipilimumab in Treating Patients With Metastatic or Recurrent Human Papilloma Virus-Related Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02877; NCI-2012-02877 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-085; PHL-085 (Other: University Health Network Princess Margaret Cancer Center P2C); 9209 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); U10CA180821 (NIH); UM1CA186705 (NIH)
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Cervical Adenocarcinoma; Cervical Squamous Cell Carcinoma; Human Papillomavirus Infection; Recurrent Cervical Carcinoma; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVB Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ipilimumab) (Experimental): Patients receive ipilimumab IV over 90 minutes. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving objective response or stable disease continue to receive maintenance therapy comprising ipilimumab IV over 90 minutes once every 12 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ipilimumab works in treating patients with human papilloma virus (HPV)-related cervical cancer that has come back or that has spread to other areas of the body. Monoclonal antibodies, such as ipilimumab, can find tumor cells and help kill them or carry tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of ipilimumab in eligible patients with recurrent or metastatic cervical cancer.

II. To assess the antitumor activity of ipilimumab in eligible patients with recurrent or metastatic cervical cancer via assessment of objective response rates (ORR).

SECONDARY OBJECTIVES:

I. To assess the antitumor activity of ipilimumab through secondary endpoints including of disease stabilization and progression free survival (PFS).

II. Assessment of antitumor activity of ipilimumab using immune-related response criteria (irRC) III. Assessment of the predictive value of baseline C-reactive protein. IV. Assess the biologic responses of exposure to ipilimumab via correlative studies involving analysis of lymphocyte subsets and assessment of cervical cancer-antigen specific T cells anti-tumor response.

V. Evaluation of archival tissue with regard to markers of immune population in correlation with clinical stage and response to treatment.

OUTLINE:

Patients receive ipilimumab intravenously (IV) over 90 minutes. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving objective response or stable disease continue to receive maintenance therapy comprising ipilimumab IV over 90 minutes once every 12 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or recurrent cervical cancer of squamous, adenocarcinoma or mixed histology type not suited to definitive localized therapy; HPV status will be confirmed for all patients following enrollment
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Previous therapy:

  * Patients may have undergone surgery and/or received definitive radiation or chemo-radiation for localized disease in the past
  * Radiation treatment with curative intent (radical chemoradiotherapy or adjuvant chemoradiotherapy) must have been completed >= 3 months prior to enrollment

    * Note: patients who completed palliative radiation therapy 2 weeks before start of ipilimumab are allowed as long as this does not affect measurable disease
  * Patients must have been exposed to platinum chemotherapy either as part of definitive chemo-radiation OR as first line systemic treatment for metastatic disease
  * Patients MAY have received up to two prior lines of systemic chemotherapy for metastatic or recurrent disease; patients with metastatic disease at first presentation MUST have received one platinum based line of chemotherapy
  * All chemotherapy must have been completed >= 4 weeks prior to enrollment with radiologic evidence of radiological disease progression
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of greater than 3 months
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin within normal institutional limits (except in Gilbert's syndrome)
* Thyroid stimulating hormone (TSH) =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine < 1.25 ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 as calculated by the Cockcroft and Gault formula
* All radiology studies must be performed =< 3 weeks prior to the start of therapy
* Subjects with treated and asymptomatic brain metastases are eligible; patients that received palliative radiation (for brain metastases) are eligible if they have been asymptomatic for at least 2 weeks with use of maintenance steroid therapy, and last received radiation at least 4 weeks prior to start of therapy
* Ability to understand and willing to sign a written informed consent document
* Ongoing prior toxicities related to previous treatments must be recovered to =< grade 1 at the time of registration (with the exception of alopecia or skin depigmentation)
* Patients are willing to undergo tumor biopsy pre-treatment (within 14 days prior to registration) and post-treatment (within the first week of cycle 2 onset); patients who consent but have tumor that is not amenable to safe biopsy will be allowed to enter the trial/continue therapy as per protocol if this has been addressed and permission is granted from the lead consortium principal investigator (PI) prior to registration continuation of treatment

Exclusion Criteria:

* Patients who have had chemotherapy < 4 weeks prior to enrollment (< 6 weeks for nitrosoureas or mitomycin C) or who had radiation therapy with curative intent < 3 months prior to enrollment (< 2 weeks for palliative radiation therapy) or those who have not recovered (=< grade 1) from adverse events related to previous treatments are excluded
* Patients with a history of prior treatment with ipilimumab or other cytotoxic T-lymphocyte antigen 4 (CTLA4) agonists or antagonists, anti-programmed death 1 (PD 1) antibody, cluster of differentiation (CD)137 agonist or other immune activating therapy such as anti-CD 40 antibody are excluded
* Patients who are receiving any other investigational agents
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and Myasthenia Gravis, multiple sclerosis)
* Patients requiring immunosuppressive agents, unless required for treating potential immune related adverse effects; steroids at their lowest effective dose in patients with radiated brain metastases is permitted
* Patients with known immune impairment who may be unable to respond to anti-CTLA 4 antibody
* Any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site or any other cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipilimumab
* Patients requiring systemic steroids are excluded; narcotics should be used with caution
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients with chronic hepatitis B or hepatitis C infections should be excluded
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ipilimumab
* Patients with active or chronic infection with human immunodeficiency virus (HIV) who have raised viral loads or uncontrolled disease are ineligible; those patients however who exhibit minimal viral loads with good control whilst on stable anti-viral regimen may be considered if they meet all other eligibility criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Oza, Principal Investigator — University Health Network Princess Margaret Cancer Center P2C
Locations (13):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Research Centre, Vancouver, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ipilimumab)
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 49 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: Cumulative count of adverse events meeting the criteria of: frequently occurring, serious and severe events of interest.
Time Frame: Up to 1 year
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
Adverse Events | 56

2. Primary Outcome: Objective Response Rate Using Response Evaluation Criteria in Solid Tumors
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
participants | 1

3. Secondary Outcome: Antitumor Activity (Partial Response, Complete Response, and Stable Disease) Using Immune-related Response Criteria (irRC)
Description: Immune-Related Complete Response (irCR): complete disappearance of all lesions for at least 4 weeks from the date of documentation of complete response. Immune-Related Partial Response (irPR): The sum of the products of the two largest perpendicular diameters of all index lesions is measured and captured as the SPD baseline. At each subsequent tumor assessment, the sum of the products of the two largest perpendicular diameters of all index lesions and of new measurable lesions are added together to provide the Immune Response Sum of Product Diameters (irSPD). A decrease, relative to baseline of the irSPD compared to the previous SPD baseline, of 50% or greater is considered an immune Partial Response (irPR). irStable Disease (irSD): does not meet criteria for irCR or irPR, in the absence of progressive disease.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
participants | 10

4. Secondary Outcome: Biologic Responses of Exposure to Ipilimumab by Analysis of Lymphocyte Subsets and Assessment of Cervical Cancer-antigen Specific T Cells Anti-tumor Response
Description: Number of Participants with Cervical Cancer-antigen Specific T Cells Anti-tumor Response
Time Frame: Up to 1 year
Population: Not collected
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Stabilization
Description: As per RECIST v1.1, stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
participants | 9

6. Secondary Outcome: Markers of Immune Population, Evaluated in Archival Tissue
Description: Evaluation of archival tissue with regard to markers of immune population in correlation with clinical stage and response to treatment
Time Frame: Baseline to 1 year after treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
participants
  PD-L1 expression negative at baseline | 20
  PD-L1 expression is 1% to 10% at baseline | 4
  PD-L1 expression is more than 10% at baseline | 4
  PD-L1 expression not available at baseline | 14
  PD-L1 expression from negative at baseline to positive after treatment | 5
  IDO expression negatve at baseline | 23
  IDO expression positive at baseline | 6
  IDO expression missing at baseline | 13

7. Secondary Outcome: Predictive Value of Baseline C-reactive Protein
Time Frame: Up to week 3 of course 4
Population: Not collected
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression Free Survival
Description: Progressive disease (PD), as per RECIST v1.1, is defined as at least a 20% increase in the sum of the diameters of target lesions and an absolute increase of at least 5mm, or the appearance of one or more new lesions. Computed using the Kaplan-Meier method.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 42
months | 2.5 [2.0 to 3.2]

ADVERSE EVENTS:
Time Frame: From treatment start and through monthly follow-up for a maximum of 1 year or until progression of disease or death (whichever occurs first).
Description: Adverse events collected as per protocol using CTCAE version 4.0
Arm/Group | Treatment (Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 25/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab) (N=42)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 3 (3)
Pelvic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ipilimumab) (N=42)
Anemia (Blood and lymphatic system disorders) | 36
Fatigue (General disorders) | 36
Lymphocyte Count Decreased (Investigations) | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 20
Abdominal Pain (Gastrointestinal disorders) | 23
HYPOALBUMINEMIA (Investigations) | 23
Anorexia (Metabolism and nutrition disorders) | 22
Nausea (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 21
Hypertension (Vascular disorders) | 15
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 19
Anxiety (Psychiatric disorders) | 14
ALKALINE PHOSPHATASE INCREASED (Investigations) | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Peripheral sensory neuropathy (Nervous system disorders) | 14
Edema Limbs (General disorders) | 15
Alanine Aminotransferase Increased (Investigations) | 14
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Aspartate Aminotransferase Increased (Investigations) | 16
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 15
Insomnia (Psychiatric disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 17
Diarrhea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 11
Cough (Ear and labyrinth disorders) | 9
Dry Mouth (Gastrointestinal disorders) | 8
Creatinine Increased (Investigations) | 12
Thromboembolic Event (Vascular disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 13
Depression (Psychiatric disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 12
Fever (General disorders) | 9
Pelvic Pain (Reproductive system and breast disorders) | 7
Sinus Tachycardia (Cardiac disorders) | 6
Hot Flashes (Vascular disorders) | 5
Neuralgia (Nervous system disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 9
Headache (Nervous system disorders) | 7
Hypothyroidism (Endocrine disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Pain (General disorders) | 5
Vaginal Discharge (Reproductive system and breast disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 5
Hydronephrosis (Renal and urinary disorders) | 4
Blurred Vision (Eye disorders) | 3
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
White Blood Cell Decreased (Investigations) | 6
Peripheral Motor Neuropathy (Nervous system disorders) | 5
Weight loss (Investigations) | 5
Urinary Tract Infection (Infections and infestations) | 5
Flatulence (Gastrointestinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Vaginal Hemorrhage (Reproductive system and breast disorders) | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 4
Urinary Frequency (Renal and urinary disorders) | 4
Hemorrhoid (Gastrointestinal disorders) | 3
Urinary Incontinence (Renal and urinary disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Acute Kidney Injury (Renal and urinary disorders) | 5
Abdominal Distension (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Lipase Increased (Investigations) | 3
Bruising (Injury, poisoning and procedural complications) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hematoma (Vascular disorders) | 4
Ascites (Gastrointestinal disorders) | 3
Localized Edema (General disorders) | 3
Paresthesia (Nervous system disorders) | 3
White Blood Cell Count Increased (Investigations) | 3
Hematuria (Renal and urinary disorders) | 4
Urinary Tract Obstruction (Renal and urinary disorders) | 3
Platelet Count Decreased (Investigations) | 3
Rectal Hemorrhage (Gastrointestinal disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
The primary limitation of the trial was the single-arm design. This was a phase 1/2 trial assessing ipilimumab monotherapy with no control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT01693783/Prot_SAP_000.pdf